CLINICAL TRIAL: NCT02035046
Title: Clinical Significance of Heterozygosity for Mutations of the SLC12A3 Gene Coding for the Thiazide Sensitive Na-Cl Cotransporter
Acronym: HEPHYGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P120111
Record Dates: First submitted 2013-12-18; First posted 2014-01-14 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Heterozygous Carriers of Gitelman Syndrome
Keywords: Gitelman; Heterozygous SLC12A3 mutation; Blood pressure; Hypokalemia
MeSH Terms: conditions — Hypokalemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study's population (Other)
  Interventions: Procedure: Samplings of blood; Procedure: Sampling of urine; Procedure: Measure of the blood pressure; Procedure: glycemia test

INTERVENTIONS:
Procedure: Samplings of blood
Procedure: Sampling of urine
Procedure: Measure of the blood pressure
Procedure: glycemia test

SUMMARY:
Gitelman syndrome is a salt wasting tubulopathy caused by mutations in the SLC12A3 gene coding for the thiazide sensitive sodium chloride cotransporter. This disease mimics the chronic treatment with thiazide diuretics and is characterized by renal hypokalemia, low to normal blood pressure, hypocalciuria and hypomagnesemia. The purpose of this study is to determine whether the heterozygous carriers present the metabolic risks and/or the benefits of this disease.

DETAILED DESCRIPTION:
Gitelman syndrome (GS), is an autosomal recessive salt wasting tubulopathy caused mainly by loss of function mutations in the SLC12A3 gene coding for the thiazide sensitive sodium-chloride cotransporter (NCC). Thus, GS mimics a chronic treatment with high doses of thiazide diuretics. NCC is expressed in the distal convoluted tubule, which is responsible for 7% of NaCl reabsorption. GS is the more frequent hereditary tubulopathie with estimated prevalence of 1/40000, which implicates that 1% of general population are heterozygous carriers (600 000 in France). Previous publications suggest that the apparently asymptomatic heterozygous carriers could present some clinical traits of GS or chronic thiazide treatment. These including: beneficial aspects (low blood pressure, low urinary calcium excretions) or metabolic risks (hypokalemia, insulin resistance). Nevertheless, these studies do not evaluate all the aspects and blood pressure was evaluated once in hospital setting. This study aims to compare home monitoring blood pressure; salt balance; potassium, glucose lipid and mineral metabolism and vascular function in 80 heterozygous carriers, 80 GS patients and 80 controls persons (without mutations in SLC12A3 gene).

ELIGIBILITY:
Gitelman syndrome patients, relatives carrying heterozygous mutations and relatives or healthy voluntarees without mutations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure evaluated by self-measurement | 3 days
  self-measurement at home, 3 times a day during 3 consecutive days

SECONDARY OUTCOMES:
Salt balance | 1 day
  Blood renin and aldosterone measurements, 24h urinary sodium and aldosterone excretion
Potassium metabolism | 1 day
  Dietary intake, blood potassium and 24 h urinary potassium excretion
Glucose and lipide metabolism | 1 day
  BMI, blood glucose, insulin, cholesterol, LDL, HDL and triglycerides.
Oral glucose tolerance test | 1 day
Mineral metabolism | 1 day
  Blood and urinary calcium, magnesium and phosphate. bone remodeling markers
Renal fonction | 1 day
  Estimated GFR, proteinuria and albuminuria
Vascular fonction evaluation | 1 day
  Pulse wave analysis and central blood pressure. Blood and urinary vascular fonction markers

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Vargas-Poussou, MD, PhD, Principal Investigator — Departement of Genetics. Assistance Publique Hôpitaux de Paris,Hôpital Européen Georges Pompidou.; Anne Blanchard, MD, PhD, Study Director — Clinical Research Center. Assistance Publique Hôpitaux de Paris, Hôpital Européen Georges Pompidou. Paris, France; Marie Essig, MD, PhD, Study Chair — Departement of Nephrology. Centre Hospitalier Universitaire. Limoges, France; Jean Philippe Haymann, MD, PhD, Study Chair — Department of Functional Investigations. Assistance Publique Hôpitaux de Paris, Hôpital Tenon, Paris, France; Ivan Tack, MD, PhD, Study Chair — Department of Functional Investigations. Centre Hospitalier Universitaire, Hôpital de Rangueil. Toulouse, France; Laurence DUBOURG, MD, PhD, Study Chair — Department of Functional Investigations. Hospices Civils de Lyon, Hôpital Edouard Herriot. Lyon, France
Locations (5):
- France (5):
  - Nephrology Department. Centre Hospitalier Universitaire, Hôpital Dupuytren, Limoges
  - Department of Functional Investigations. Hospices Civils de Lyon, Hôpital Edouard Herriot., Lyon
  - Department of Functional Investigations. Assistance Publique Hôpitaux de Paris, Hôpital Tenon, Paris
  - Clinical Research Center. Assistance Publique Hôpitaux de Paris, Hôpital Européen Georges Pompidou., Paris
  - Department of Functional Investigations. Centre Hospitalier Universitaire, Hôpital de Rangueil., Toulouse

REFERENCES:
- [Background] Tago N, Kokubo Y, Inamoto N, Naraba H, Tomoike H, Iwai N. A high prevalence of Gitelman's syndrome mutations in Japanese. Hypertens Res. 2004 May;27(5):327-31. doi: 10.1291/hypres.27.327. PMID 15198479
- [Background] Fava C, Montagnana M, Rosberg L, Burri P, Almgren P, Jonsson A, Wanby P, Lippi G, Minuz P, Hulthen LU, Aurell M, Melander O. Subjects heterozygous for genetic loss of function of the thiazide-sensitive cotransporter have reduced blood pressure. Hum Mol Genet. 2008 Feb 1;17(3):413-8. doi: 10.1093/hmg/ddm318. Epub 2007 Nov 1. PMID 17981812
- [Background] Ji W, Foo JN, O'Roak BJ, Zhao H, Larson MG, Simon DB, Newton-Cheh C, State MW, Levy D, Lifton RP. Rare independent mutations in renal salt handling genes contribute to blood pressure variation. Nat Genet. 2008 May;40(5):592-599. doi: 10.1038/ng.118. Epub 2008 Apr 6. PMID 18391953
- [Background] Hsu YJ, Yang SS, Chu NF, Sytwu HK, Cheng CJ, Lin SH. Heterozygous mutations of the sodium chloride cotransporter in Chinese children: prevalence and association with blood pressure. Nephrol Dial Transplant. 2009 Apr;24(4):1170-5. doi: 10.1093/ndt/gfn619. Epub 2008 Nov 25. PMID 19033254
- [Background] Ren H, Qin L, Wang W, Ma J, Zhang W, Shen PY, Shi H, Li X, Chen N. Abnormal glucose metabolism and insulin sensitivity in Chinese patients with Gitelman syndrome. Am J Nephrol. 2013;37(2):152-7. doi: 10.1159/000346708. Epub 2013 Jan 31. PMID 23392128
- [Background] Cruz DN, Simon DB, Nelson-Williams C, Farhi A, Finberg K, Burleson L, Gill JR, Lifton RP. Mutations in the Na-Cl cotransporter reduce blood pressure in humans. Hypertension. 2001 Jun;37(6):1458-64. doi: 10.1161/01.hyp.37.6.1458. PMID 11408395